CLINICAL TRIAL: NCT00937638
Title: BOLD (Beef in an Optimal Lean Diet) Effects on Established and Emerging Cardiovascular Disease (CVD) Risk Factors: Effects on Metabolic Syndrome (BOLD-X)
Brief Title: Beef in an Optimal Lean Diet (BOLD) Effects on Metabolic Syndrome
Acronym: BOLD-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKE BOLD-X
Record Dates: First submitted 2009-06-18; First posted 2009-07-13 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome; Cardiovascular Disease
Keywords: Metabolic syndrome; Lean Beef; CVD
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases | interventions — Diet, Fat-Restricted; Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modified-DASH Diet (Experimental)
  Interventions: Dietary Supplement: Modified DASH Diet
- BOLD diet (Experimental)
  Interventions: Dietary Supplement: BOLD Diet
- BOLD-X (Experimental)
  Interventions: Dietary Supplement: BOLD-X Diet

INTERVENTIONS:
Dietary Supplement: BOLD Diet — Low-fat, high fruit and vegetable diet that includes lean beef (5oz/day)
  Other Names: Low fat, Step II diet
  Arms: BOLD diet
Dietary Supplement: BOLD-X Diet — Low-fat, moderate-high protein diet (BOLD+) that is higher in total protein (from mixed sources including lean beef, 7oz/day) than the BOLD diet. Also high in fruits and vegetables
  Other Names: Low fat, moderate protein
  Arms: BOLD-X
Dietary Supplement: Modified DASH Diet — Low-fat, high fruit and vegetable diet which has become the Gold Standard for the management of cardiovascular disease (CVD) risk factors and metabolic syndrome
  Other Names: DASH diet
  Arms: Modified-DASH Diet

SUMMARY:
The proposed research will provide important information about the role of 2 intervention diets that provide different amounts of lean beef and meet current nutrient recommendations for the treatment of Metabolic Syndrome (MetSyn), a chronic disease that is still increasing in prevalence at alarming rates. The experimental and diet designs will enable us to evaluate lifestyle interventions for MetSyn for persons who maintain weight, lose weight and maintain their weight loss, as is currently recommended in clinical practice. Importantly, the investigators will compare a diet high in lean beef (5 oz/day) which is compositionally similar (i.e., energy and nutrients) to the modified-DASH diet, a low beef diet which has become the Gold Standard for the management of cardiovascular disease (CVD) risk factors, including MetSyn. In addition, the investigators also will evaluate a moderate-high protein diet (BOLD+) that is higher in total protein (from mixed sources including lean beef, 7oz/day) than the BOLD diet, on CVD risk factors in persons with MetSyn. A follow-up study was conducted to assess dietary compliance in a sub-sample of the population at 12-months; participants were not informed of this end-point and additional consent was obtained.

Hypotheses:

1. Healthful isocaloric diets that include lean beef as the primary source of protein (BOLD diet) with average (18%; BOLD) or moderate-high (28%; BOLD+) total protein intake will show similar or greater reductions in CVD risk, respectively when compared to a modified-DASH diet.
2. A healthful weight-loss diet, including lean beef as the primary source of protein in a high-moderate protein diet (BOLD+ diet), plus regular exercise (BOLD+ + ex) will reduce body weight equal to that of a BOLD + ex and DASH + ex intervention, but may improve CV risk factors (such as BP and TG), and therefore reduce the prevalence of MetSyn more than a BOLD + ex and DASH + ex intervention.
3. The BOLD diet will be more effective than the modified-DASH diet, and the BOLD+ diet more effective than the BOLD diet in maintaining the CVD benefits attained during phases 1 and 2. Dietary adherence will be better on the BOLD and BOLD + diets compared with the modified DASH diet.

ELIGIBILITY:
Inclusion Criteria:

* (BMI 27-42 kg/m2)
* Three or more of the following risk factors (defined as having MetSyn):

  * abdominal obesity [waist circumference > 102 cm (40 inches) in men and > 88 cm (35 inches) in women],
  * elevated blood glucose [> 110mg/dl (6.1 mmol/L)]
  * elevated TG [>150 mg/dl (1.7 mmol/L)]
  * low HDL-C [<40 mg/dl (1.03 mmol/L) in men and <50 mg/dL (1.29 mmol/l) in women]
  * hypertension (Systolic Blood Pressure > 130 mmHg or Diastolic Blood Pressure > 85 mmHg)*

    * BP medication accepted if BP stable and less than 160/100mm Hg

Exclusion Criteria:

* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease (unless controlled on medication)
* Lactation, pregnancy, or desire to become pregnant during the study
* Intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, and phytoestrogens, stanol/sterol supplemented foods)
* High alcohol consumption (≥ 14 drinks/week)
* Participation in regular physical activity (> 1 formal session/week)
* Lipid or glucose lowering medication

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Criteria for Metabolic Syndrome: central obesity (weight, waist circumference, abdominal obesity), TG, HDL-C, glucose and BP | 2 weeks
Criteria for Metabolic Syndrome: central obesity (weight, waist circumference, abdominal obesity), TG, HDL-C, glucose and BP | 7 weeks
Criteria for Metabolic Syndrome: central obesity (weight, waist circumference, abdominal obesity), TG, HDL-C, glucose and BP | 13 weeks
Criteria for Metabolic Syndrome: central obesity (weight, waist circumference, abdominal obesity), TG, HDL-C, glucose and BP | 24 weeks

SECONDARY OUTCOMES:
Vascular endothelial function measured by endo-PAT | 2 weeks
Lipids and lipoproteins | 2 weeks
Inflammatory markers | 2 weeks
Vascular endothelial function measured by endo-PAT | 7 weeks
Vascular endothelial function measured by endo-PAT | 13 weeks
Vascular endothelial function measured by endo-PAT | 24 weeks
Lipids and lipoproteins | 7 weeks
Lipids and lipoproteins | 13 weeks
Lipids and lipoproteins | 24 weeks
Inflammatory markers | 7 weeks
Inflammatory markers | 13 weeks
Inflammatory markers | 24 weeks
Dietary analysis | 52 weeks
  macro-and micronutrients
Criteria for Metabolic Syndrome: central obesity (weight, waist circumference) TG, HDL-C, glucose and BP | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Hill AM, Harris Jackson KA, Roussell MA, West SG, Kris-Etherton PM. Type and amount of dietary protein in the treatment of metabolic syndrome: a randomized controlled trial. Am J Clin Nutr. 2015 Oct;102(4):757-70. doi: 10.3945/ajcn.114.104026. Epub 2015 Sep 9. PMID 26354540